CLINICAL TRIAL: NCT01267890
Title: Health Service Administration China Medical University (Chih-Jaan Tai)
Brief Title: The Conflicts of Ethics and Law on Patient's Surrogate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Chih-Jaan Tai, China Medical University Hospital
Other Study IDs: CMU-DMR99-IRB-254
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Physician's Role
Keywords: ethics; law; surrogate; conflict

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a prospective cross-sectional survey study. The investigators developed self-administrated questionnaire and recruit 120 physicians in two hospitals and 60 lawyers from some law firms to this study.

To realize and compare the opinions of physicians and lawyers about controversial decision-making of surrogate.

DETAILED DESCRIPTION:
This study provides three real scenarios regarding dilemma between ethics and law when patient's surrogate may not represent patient's best interest：1. Parents ask physician resect their mentally handicapped daughter's uterus. 2. A son refuse physician's suggestion of surgical treatment for his mother, instead, wishes donating his mother's kidney to his son. 3. A mother decides to give up treatment for her son's head injury because of his rebel behavior before.

T-test, ANOVA and Logistic Regression will be used to analyze in this study.

ELIGIBILITY:
Inclusion Criteria:

* resident
* visiting Staff
* chief resident

Exclusion Criteria:

* intern
* clerk

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 120 physicians in two hospitals
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-05 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan